CLINICAL TRIAL: NCT00666276
Title: Drug Use Investigation Of Zyvox (Linezolid) (Regulatory Post Marketing Commitment Plan)
Status: Completed | Type: Observational
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Other Study IDs: A5951142
Record Dates: First submitted 2008-04-22; First posted 2008-04-24 (Estimated); Results first posted 2012-07-02 (Estimated); Last update posted 2012-07-02 (Estimated); Status verified 2012-05

CONDITIONS: Staphylococcal Infections
MeSH Terms: conditions — Staphylococcal Infections | interventions — Linezolid

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- linezolid (Zyvox): Patients taking Linezolid.
  Interventions: Drug: linezolid (Zyvox)

INTERVENTIONS:
Drug: linezolid (Zyvox) — Zyvox Tablets 600mg, Zyvox Injection 600mg Dosage, Frequency: According to Japanese Package Insert, In adults, administer usually 600mg of linezolid twice daily (q 12 hours) for a total daily dose of 1200 mg.
  Duration: According to the protocol of A5951142, the duration of the investigation for findings regarding safety and efficacy of a patient is from the first drug administration to the 8 weeks after the first administration.

SUMMARY:
Drug use investigation of Zyvox for patients with Methicillin-resistant Staphylococcus aureus (MRSA) infection disease.

The objective of this surveillance is to collect information about 1) adverse drug reaction not expected from the Package Insert (unknown adverse drug reaction), 2) the incidence of adverse drug reactions in this surveillance, and 3)factors considered to affect the safety and/or efficacy of this drug.

DETAILED DESCRIPTION:
All the patients whom an investigator prescribes the first Linezolid should be registered consecutively until the number of subjects reaches target number in order to extract patients enrolled into the investigation at random.

ELIGIBILITY:
Inclusion Criteria:

* Patients need to be administered Linezolid in order to be enrolled in the surveillance.

Exclusion Criteria:

* Patients not administered Linezolid.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The patients whom an investigator involving A5951142 prescribes the Linezolid.
Sampling Method: Probability Sample
Enrollment: 1004 (Actual)
Dates: Start 2007-02; Primary Completion 2011-04 (Actual); Study Completion 2011-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This was an open label, prospective, multi-center non-interventional cohort study.
Groups:
- Linezolid: Participants who have been treated with Linezolid.
Period: Overall Study
Arm/Group | Linezolid
Started | 1004
Completed | 970
Not Completed | 34
Not completed — Protocol Violation | 34

BASELINE CHARACTERISTICS:
Arm/Group | Linezolid
Number analyzed (Participants) | 970
Age, Customized [Number; unit: participants]
  <65 years | 282
  >=65 years | 688
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 308
  Male | 662
Target disease [Number; unit: participants] — The physician in charge of the study made the diagnosis of Target disease based on symptoms.
  participants
    Sepsis | 192
    Deep-seated skin infection | 33
    Secondary infection in injury, Burn and operative | 136
    Pneumonia | 377
    Multiple infection | 141
    Other | 91
Target disease Severity [Number; unit: participants]
  Mild | 68
  Moderate | 455
  Severe | 447
Complications [Number; unit: participants] — Complications is the patient's current experiences with illnesses, operations, injuries and treatments. The physician of this survey made the diagnosis. (e.g. hypertension, diabetes, etc.)
  participants
    Present | 897
    Absent | 73

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Adverse Drug Reaction Not Expected From the Japanese Package Insert.
Description: The adverse drug reaction that have not been listed in Japanese package insert.
Time Frame: Baseline to 8 weeks
Population: Safety analysis population consists of the participants that satisfy the inclusion and exclusion conditions and in whom administration of this drug was confirmed.
Measure: Number; unit: participants
Arm/Group | Linezolid
Number analyzed (Participants) | 970
participants
  Superinfection | 1
  Sepsis | 1
  Thrombocytopenia | 1
  Lactic acidosis | 1
  Agitation | 1
  Deep vein thrombosis | 1
  Hyperbilirubinaemia | 1
  Antithrombin III decreased | 1
  Blood chloride increased | 1
  Blood sodium increased | 1

2. Primary Outcome: Number of Participants With Adverse Drug Reactions(ADRs).
Description: All observed or volunteered adverse events and the investigator's opinion of the causal relationship to the study treatment were reported. Adverse Drug Reactions were evaluated in company with the causal relationship to the investigational product.
Time Frame: 8 weeks
Population: as for outcome 1
Measure: Number; unit: participants
Arm/Group | Linezolid
Number analyzed (Participants) | 970
participants | 163

3. Primary Outcome: Factors Considered to Affect the Safety of Linezolid - Gender.
Description: Number of participants with adverse drug reaction to determine whether male or female is significant risk factor.
Time Frame: 8 weeks
Population: as for outcome 1
Measure: Number; unit: participants
Groups:
- Linezolid-male: Male participants who have been treated with Linezolid.
- Linezolid-female: Female participants who have been treated with Linezolid.
Arm/Group | Linezolid-male | Linezolid-female
Number analyzed (Participants) | 662 | 308
participants | 109 | 54
Statistical Analysis 1: Comparison: Linezolid-male vs Linezolid-female; The risk factor tested was "Gender". The null hypothesis is there is no difference between "males and females" in the incidence rate of ADRs; Test type: Superiority or Other; p = 0.712, Fisher Exact

4. Primary Outcome: Factors Considered to Affect the Safety of Linezolid - Age
Description: Number of participants with adverse drug reaction to determine whether over 65 or less than 65 is significant risk factor.
Time Frame: 8 weeks
Population: as for outcome 1
Measure: Number; unit: participants
Groups:
- Linezolid-over 65: Participants with over 65 years old who have been treated with Linezolid.
- Linezolid-less Than 65: Participants with less than 65 years old who have been treated with Linezolid.
Arm/Group | Linezolid-over 65 | Linezolid-less Than 65
Number analyzed (Participants) | 688 | 282
participants | 122 | 41
Statistical Analysis 1: Comparison: Linezolid-over 65; The risk factor tested was "Age". The null hypothesis is there is no difference between "over 65 and less than 65" in the incidence rate of ADRs; Test type: Superiority or Other; p = 0.257, Fisher Exact

5. Primary Outcome: Factors Considered to Affect the Safety of Linezolid - Hepatic Dysfunctions.
Description: Number of participants with or without Hepatic dysfunctions with adverse drug reaction to determine whether with or without is significant risk factor.
Time Frame: 8 weeks
Population: as for outcome 1
Measure: Number; unit: participants
Groups:
- Linezolid-without Hepatic Dysfunctions: Participants with or without Hepatic dysfunctions who have been treated with Linezolid.
- Linezolid- With Hepatic Dysfunctions: Participants with Hepatic dysfunctions who have been treated with Linezolid.
Arm/Group | Linezolid-without Hepatic Dysfunctions | Linezolid- With Hepatic Dysfunctions
Number analyzed (Participants) | 856 | 114
participants | 137 | 26
Statistical Analysis 1: Comparison: Linezolid-without Hepatic Dysfunctions vs Linezolid- With Hepatic Dysfunctions; The risk factor tested was "Hepatic dysfunctions". The null hypothesis is there is no difference between "with Hepatic dysfunction and without Hepatic dysfunction" in the incidence rate of ADRs; Test type: Superiority or Other; p = 0.082, Fisher Exact

6. Primary Outcome: Factors Considered to Affect the Safety of Linezolid - Renal Dysfunctions.
Description: Number of participants with or without Renal dysfunctions with adverse drug reaction to determine whether with or without is significant risk factor.
Time Frame: 8 weeks
Population: as for outcome 1
Measure: Number; unit: participants
Groups:
- Linezolid Without Renal Dysfunctions: Participants without Renal dysfunctions who have been treated with Linezolid.
- Linezolid- With Renal Dysfunctions: Participants with Renal dysfunctions who have been treated with Linezolid.
Arm/Group | Linezolid Without Renal Dysfunctions | Linezolid- With Renal Dysfunctions
Number analyzed (Participants) | 765 | 205
participants | 125 | 38
Statistical Analysis 1: Comparison: Linezolid Without Renal Dysfunctions vs Linezolid- With Renal Dysfunctions; The risk factor tested was "Renal dysfunctions". The null hypothesis is there is no difference between "with Renal dysfunction and without Renal dysfunction" in the incidence rate of ADRs; Test type: Superiority or Other; p = 0.462, Fisher Exact

7. Primary Outcome: Factors Considered to Affect the Safety of Linezolid - Duration of Drug Administration.
Description: Number of participants with Duration of drug administration as over 15 days or less than 15 days with adverse drug reaction to determine whether over 15 days or less than 15 days is significant risk factor.
Time Frame: 8 weeks
Population: as for outcome 1
Measure: Number; unit: participants
Groups:
- Linezolid-administrated Over 15 Days: Participants who have been treated with Linezolid.with Duration of drug administration over 15 days
- Linezolid-administrated Less Than 15 Days: Participants with who have been treated with Linezolid.with Duration of drug administration less than 15 days
Arm/Group | Linezolid-administrated Over 15 Days | Linezolid-administrated Less Than 15 Days
Number analyzed (Participants) | 203 | 767
participants | 53 | 110
Statistical Analysis 1: Comparison: Linezolid-administrated Over 15 Days vs Linezolid-administrated Less Than 15 Days; The risk factor tested was "Duration of drug administration". The null hypothesis is there is no difference between "over 15 days and less than 15 days" in the incidence rate of ADRs; Test type: Superiority or Other; p < 0.001, Fisher Exact

8. Primary Outcome: Factors Considered to Affect the Safety of Linezolid - Route of Administration.
Description: Number of participants Route of administration as by oral,injection or oral from injection with adverse drug reaction to determine whether oral, injection or switch is significant risk factor.
Time Frame: 8 weeks
Population: as for outcome 1
Measure: Number; unit: participants
Groups:
- Linezolid-oral: Participants with who have been orally treated with Linezolid.
- Linezolid-injection: Participants with who have been treated with Linezolid by injection.
- Linezolid-oral From Injection: Participants with who have been treated with Linezolid by orally from injection .
Arm/Group | Linezolid-oral | Linezolid-injection | Linezolid-oral From Injection
Number analyzed (Participants) | 132 | 768 | 70
participants | 29 | 116 | 18
Statistical Analysis 1: Comparison: Linezolid-oral vs Linezolid-injection vs Linezolid-oral From Injection; The risk factor tested was "Route of administration". The null hypothesis is there is no difference between "oral, injection and switch" in the incidence rate of ADRs; Test type: Superiority or Other; p = 0.018, Fisher Exact

9. Primary Outcome: Factors Considered to Affect the Safety of Linezolid - Weight.
Description: Number of participants Weight as over 40kg or less than 40kg with adverse drug reaction to determine whether over 40kg or less than 40kg Weight is significant risk factor.
Time Frame: 8 weeks
Population: as for outcome 1
Measure: Number; unit: participants
Groups:
- Linezolid -Over 40kg: Participants over 40kg who have been treated with Linezolid.
- Linezolid -Less Than 40kg: Participants less than 40kg who have been treated with Linezolid.
Arm/Group | Linezolid -Over 40kg | Linezolid -Less Than 40kg
Number analyzed (Participants) | 651 | 96
participants | 108 | 20
Statistical Analysis 1: Comparison: Linezolid -Over 40kg vs Linezolid -Less Than 40kg; The risk factor tested was "Weight". The null hypothesis is there is no difference between "over 40kg and less than 40kg" in the incidence rate of ADRs; Test type: Superiority or Other; p = 0.311, Fisher Exact

10. Primary Outcome: Factors Considered to Affect the Safety of Linezolid - Concomitant Drugs.
Description: Number of participants with or without Concomitant drugs with adverse drug reaction to determine whether with or without is significant risk factor.
Time Frame: 8 weeks
Population: as for outcome 1
Measure: Number; unit: participants
Groups:
- Linezolid-without Concomitant Drugs: Participants without Concomitant drugs who have been treated with Linezolid.
- Linezolid-with Concomitant Drugs: Participants with Concomitant drugs who have been treated with Linezolid.
Arm/Group | Linezolid-without Concomitant Drugs | Linezolid-with Concomitant Drugs
Number analyzed (Participants) | 97 | 873
participants | 9 | 154
Statistical Analysis 1: Comparison: Linezolid-without Concomitant Drugs vs Linezolid-with Concomitant Drugs; The risk factor tested was "Concomitant drugs". The null hypothesis is there is no difference between "with Concomitant drug and without Concomitant drug" in the incidence rate of ADRs; Test type: Superiority or Other; p = 0.044, Fisher Exact

11. Primary Outcome: Factors Considered to Affect the Safety of Linezolid - Non-drug Therapies.
Description: Number of participants with or without Non-drug therapies with adverse drug reaction to determine whether with or without is significant risk factor.
Time Frame: 8 weeks
Population: as for outcome 1
Measure: Number; unit: participants
Groups:
- Linezolid-without Non-drug Therapies: Participants without Non-drug therapies who have been treated with Linezolid.
- Linezolid-with Non-drug Therapies: Participants with Non-drug therapies who have been treated with Linezolid.
Arm/Group | Linezolid-without Non-drug Therapies | Linezolid-with Non-drug Therapies
Number analyzed (Participants) | 610 | 360
participants | 87 | 76
Statistical Analysis 1: Comparison: Linezolid-without Non-drug Therapies vs Linezolid-with Non-drug Therapies; The risk factor tested was "Non-drug therapies". The null hypothesis is there is no difference between "with Non-drug therapies and without Non-drug therapies" in the incidence rate of ADRs; Test type: Superiority or Other; p = 0.008, Fisher Exact

ADVERSE EVENTS:
Description: The same event may appear as both an AE and a SAE. However, what is presented are distinct events. An event may be categorized as serious in one subject and as nonserious in another subject, or one subject may have experienced both a serious and nonserious event during the study.
Arm/Group | Linezolid
Serious Adverse Events (participants affected / at risk) | 50/970
Other Adverse Events (participants affected / at risk) | 163/970
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Linezolid (N=970)
Platelet count decreased (Investigations) | 23 (23)
Thrombocytopenia (Blood and lymphatic system disorders) | 10 (10)
Anaemia (Blood and lymphatic system disorders) | 7 (7)
Bone marrow failure (Blood and lymphatic system disorders) | 3 (3)
Pancytopenia (Blood and lymphatic system disorders) | 3 (3)
Haemoglobin decreased (Investigations) | 3 (3)
White blood cell count decreased (Investigations) | 3 (3)
Superinfection (Infections and infestations) | 2 (2)
Haematocrit decreased (Investigations) | 2 (2)
Red blood cell count decreased (Investigations) | 2 (2)
Sepsis (Infections and infestations) | 1 (1)
Lactic acidosis (Metabolism and nutrition disorders) | 1 (1)
Deep vein thrombosis (Vascular disorders) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 1 (1)
Hyperbilirubinaemia (Hepatobiliary disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Linezolid (N=970)
Platelet count decreased (Investigations) | 78 (78)
Anaemia (Blood and lymphatic system disorders) | 31 (31)
Thrombocytopenia (Blood and lymphatic system disorders) | 26 (26)
White blood cell count decreased (Investigations) | 12 (12)
Bone marrow failure (Blood and lymphatic system disorders) | 8 (8)
Hepatic function abnormal (Hepatobiliary disorders) | 6 (6)
Superinfection (Infections and infestations) | 5 (5)
Diarrhoea (Gastrointestinal disorders) | 5 (5)
Pancytopenia (Blood and lymphatic system disorders) | 4 (4)
Rash (Skin and subcutaneous tissue disorders) | 4 (4)
Drug eruption (Skin and subcutaneous tissue disorders) | 4 (4)
Haemoglobin decreased (Investigations) | 4 (4)
Decreased appetite (Metabolism and nutrition disorders) | 3 (3)
Hyponatraemia (Metabolism and nutrition disorders) | 3 (3)
Red blood cell count decreased (Investigations) | 3 (3)
Hyperkalaemia (Metabolism and nutrition disorders) | 2 (2)
Hypochloraemia (Metabolism and nutrition disorders) | 2 (2)
Haematocrit decreased (Investigations) | 2 (2)
Blood bilirubin increased (Investigations) | 2 (2)
Pneumonia klebsiella (Infections and infestations) | 1 (1)
Pseudomonas infection (Infections and infestations) | 1 (1)
Sepsis (Infections and infestations) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 1 (1)
Lactic acidosis (Metabolism and nutrition disorders) | 1 (1)
Agitation (Nervous system disorders) | 1 (1)
Deep vein thrombosis (Vascular disorders) | 1 (1)
Reflux oesophagitis (Gastrointestinal disorders) | 1 (1)
Enterocolitis (Gastrointestinal disorders) | 1 (1)
Vomiting (Gastrointestinal disorders) | 1 (1)
Liver disorder (Hepatobiliary disorders) | 1 (1)
Hyperbilirubinaemia (Hepatobiliary disorders) | 1 (1)
Aspartate aminotransferase increased (Investigations) | 1 (1)
Alanine aminotransferase increased (Investigations) | 1 (1)
Antithrombin III decreased (Investigations) | 1 (1)
Liver function test abnormal (Investigations) | 1 (1)
Blood chloride increased (Investigations) | 1 (1)
Blood sodium increased (Investigations) | 1 (1)
Blood glucose increased (Investigations) | 1 (1)
Blood urea increased (Investigations) | 1 (1)
White blood cell count increased (Investigations) | 1 (1)
Reticulocyte count decreased (Investigations) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.